CLINICAL TRIAL: NCT04911946
Title: Evaluation of the Management of Patients With Osteoporotic Fractures by Orthopedics Residents: an Observational Cross-sectional Study
Brief Title: Training of Orthopedic Residents in OP Treatment
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1445; 38248820.1.0000.0068 (Other: CAAE)
Record Dates: First submitted 2021-05-06; First posted 2021-06-03 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-05

CONDITIONS: Osteoporotic Fractures
Keywords: Osteoporotic fractures; Secondary prevention; Brazil; Orthopedics; Medical professionals; Knowledge Gap; Osteoporosis treatment
MeSH Terms: conditions — Osteoporotic Fractures | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- R1: Resident of the first year of orthopedics and traumatology at IOT-HC-FMUSP.
  Interventions: Other: Questionnaire
- R2: Resident of the second year of orthopedics and traumatology at IOT-HC-FMUSP.
  Interventions: Other: Questionnaire
- R3: Resident of the third year of orthopedics and traumatology at IOT-HC-FMUSP.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — After signing the informed consent form agreeing to participate in the study, the participants answered the questionnaire about diagnostic and therapeutic questions related to a clinical case of osteoporotic fracture in 4 scenarios: the initial care in the emergency room, at the time of discharge from hospital, during their outpatient return in 3 and 6 months.

SUMMARY:
Objective: To assess whether residents (R1, R2 or R3 according to the year of residency) of an orthopedic tertiary service, investigate, treat and / or refer the patient with an osteoporotic fracture to treat osteoporosis (OP) and whether this learning is improved over the years of residence.

Methods: Residents answered diagnostic and therapeutic questions related to a clinical case of osteoporotic fracture (OF) in 4 scenarios, which were the initial care in the emergency room, at the time of discharge from hospital, during their outpatient return in 3 and 6 months. Answers were compared between years of residence.

ELIGIBILITY:
Inclusion Criteria:

* Physicians enrolled in the medical residency program in orthopedics and traumatology at IOT-HC-FMUSP.

Exclusion Criteria:

* Abandonment of the medical residency program in orthopedics and traumatology at IOT-HC-FMUSP.
* Withdrawal from the medical residency program in orthopedics and traumatology at the IOT-HC-FMUSP for a period of more than 120 days.
* Expulsion from the medical residency program in orthopedics and traumatology at IOT-HC-FMUSP.
* Transfer of the medical residency program in orthopedics and traumatology from IOT-HC-FMUSP to another institution.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians enrolled in the medical residency program in orthopedics and traumatology at IOT-HC-FMUSP.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Secondary prevention of osteoporotic fracture | through study completion, an average of 1 month
  Number of residents investigating and treating osteoporosis in an appropriate manner

SECONDARY OUTCOMES:
Patient referral to secondary prevention of osteoporotic fracture | through study completion, an average of 1 month
  Number of residents that does not start osteoporosis treatment but refer the patient to another professional to conduct the case.
Change the proficiency of secondary prevention with increasing graduation in the residency program | through study completion, an average of 1 month
  Increase the number of residents who adequately treat osteoporosis categorized by year of graduation

CONTACTS AND LOCATIONS:
Overall Officials: Marcia U Rezende, PhD MD, Principal Investigator — Instituto de Ortopedia e Traumatologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided